CLINICAL TRIAL: NCT06078995
Title: Tenecteplase Thrombolytic Therapy for Acute Ischemic Stroke in China a Real-world, Multicenter, Retrospective, Controlled Study
Brief Title: Tenecteplase Thrombolytic Therapy for Acute Ischemic Stroke in China
Acronym: TTT-AIS CHINA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Keshiketeng Banner Traditional Chinese Medicine Mongolian Medicine Hospitalorem Ipsum (Unknown); Nanshi Hospital of Nanyang (Unknown); First Affiliated Hospital of Ningbo University (Network); Jilin Liuhe Hospital (Unknown); Shenyang Fifth People's hospital (Unknown); Shanghai East Hospita (Unknown); Shanghai 10th People's Hospital (Other); Shanghai Fifth People's Hospital (Unknown); Shanghai Pudong Gongli hospital (Unknown); Shanghai Neuromedical Center (Unknown); Shanghai Fourth People's Hospital (Unknown); Shanghai Pudong People's Hospital (Unknown); Shanghai Putuo District Center Hospital (Other); Shenyang Fushun general hospital of mining bureau (Unknown); Yantai Affliated Hosiptal of Binzhou Medical University (Unknown); Shanghai Ninth People's Hospital Huangpu Branch (Unknown); Shanghai Deji Hospital (Unknown); Ruijin Hospital Luwan Branch (Other)
Responsible Party: Principal Investigator, Qiang Dong, Professor, Huashan Hospital
Other Study IDs: 20230726
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Stroke
Keywords: intravenous thrombolysis; Tenecteplase
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tenecteplase: acute ischemic stroke patients who receive intravenous thrombolysis with tenecteplase
  Interventions: Drug: Tenecteplase
- alteplase: acute ischemic stroke patients who receive intravenous thrombolysis with alteplase
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Tenecteplase — Thrombolysis wtih rhTNK-tPA
  Other Names: rhTNK-tPA
  Groups: Tenecteplase
Drug: Alteplase — Thrombolysis wtih rt-PA
  Other Names: rt-PA
  Groups: alteplase

SUMMARY:
The objective of the study is to investigate the effectiveness and safety of rhTNK-tPA in acute ischemic stroke patients within 4.5 hours of symptom onset in a real-world clinical setting.

DETAILED DESCRIPTION:
Recombinant human tenecteplase tissue-type plasminogen activator (rhTNK-tPA) has the logistic advantage of a single bolus infusion over recombinant tissue plasminogen activator (rt-PA) which needs a 1-hour infusion. The non-inferiority of rhTNK-tPA compared to rt-PA was proved by two recent randomized controlled clinical trials but the evidence is lacking regarding the real-world effectiveness and safety of rhTNK-tPA.

This is a multi-center, observational, retrospective study that enrolled acute ischemic stroke patients treated with rhTNK-tPA thrombolysis in China.

ELIGIBILITY:
Inclusion Criteria:

* all acute ischaemic stroke patients who met eligibility for thrombolysis with intravenous alteplase or TNK and presenting within 4·5 hours of symptom onset.

Exclusion Criteria:

* variables with a missing rate > 40%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute ischemic stroke patients treated with rhTNK-tPA or rt-PA in China.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with symptomatic intracranial hemorrhage within 36 hours | 36 hours
  Clinical deterioration or neurological decline causing an increase in NIHSS score of ≥4 points due to intracranial hemorrhage confirmed by brain imaging

SECONDARY OUTCOMES:
90 days mRS 0-1 | at 90±7 days
  modified Rankin Scale score measures degree of disability/dependence after a stroke. Patients are graded on the scale of 0-6, with higher scores indicating worse functional outcome. 0 means no symptoms, 6 means death.
90 days mRS shift | at 90±7 days
  a shift analysis of the distribution of modified Rankin Scale score which measures degree of disability/dependence after a stroke. Patients are graded on the scale of 0-6, with higher scores indicating worse functional outcome. 0 means no symptoms, 6 means death.
discharge mRS | at discharge (up to 30 days)
  modified Rankin Scale score measures degree of disability/dependence after a stroke. Patients are graded on the scale of 0-6, with higher scores indicating worse functional outcome. 0 means no symptoms, 6 means death.
24 hours NIHSS score | at 24 hours after receiving thrombolysis
  The NIH Stroke Scale/Score (NIHSS) quantifies stroke severity based on weighted evaluation findings. Scores range from 0 to 42, with higher scores indicating greater severity.
discharge NIHSS score | at discharge (up to 30 days)
  The NIH Stroke Scale/Score (NIHSS) quantifies stroke severity based on weighted evaluation findings. Scores range from 0 to 42, with higher scores indicating greater severity.
Rate of patients with any systematic bleeding | during hospital stay (up to 30 days)
  Rate of patients with any systematic bleeding requiring blood infusion during hospital stay reflecting short term safety outcome
Rate of patients with 90 days mortality | at 90±7 days
  Rate of patients with all-cause mortality within 90 days reflecting safety outcome
Rate of patients with any intracranial hemorrhage | during hospital stay (up to 30 days)
  Rate of patients with any intracranial hemorrhage without significant neurological deterioration on the brain imaging reflecting short term safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Dong, Principal Investigator — Huashan Hospital
Locations (1):
- Xin Chen, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided